CLINICAL TRIAL: NCT04628728
Title: Possibilities and Measures to Improve Health Literacy
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: EK_NR_31-366 ex 18/19
Record Dates: First submitted 2020-11-04; First posted 2020-11-13 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Health Care Utilization; Medication Compliance; Information Seeking Behavior
MeSH Terms: conditions — Patient Acceptance of Health Care; Medication Adherence; Information Seeking Behavior

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Current referral letters: One letter will be chosen from the selection of current referral letters (of average quality according to the results of the study mentioned above). Any data that would allow identification of the respective patient (i.e. name, date of birth, social insurance number, address) will be anonymised (not blackened in order not to disturb fluent reading).
  Interventions: Other: Survey based on questionnaire (self-designed)
- New referral letters: The other one will be a corrected version of the first letter according to the ELGA (Elektronische Gesundheitsakte) requirements and the identified needs of patients and stakeholders (see Previous Work 1).
  Interventions: Other: Survey based on questionnaire (self-designed)

INTERVENTIONS:
Other: Survey based on questionnaire (self-designed) — Participants are handed a questionnaire to asses comprehension of medical content provided in the referral letters.

SUMMARY:
Health literacy describes one's capability to understand and implement health information in daily practice. Hospital referral letters remain a main information tool for patients as well as physicians with information about therapeutic measures done during hospital stay as well as recommendations on drug intake, further therapies or diagnostics to be done after hospital discharge.

With increasing medical knowledge, hospital referral letters have become more difficult to understand for patients and stakeholders alike. The aim of this study is to develop a patient-friendly referral letter that is easier to understand while transporting the same amount of information for patients as well as stakeholders.

DETAILED DESCRIPTION:
During the last decades healthcare systems had to face new challenges in patient care: Along with increasing life expectancy and better treatment options for many diseases also the amount of chronically ill elderly patients increased. Much is expected of this particular patient group regarding self-management and comprehension of their medical condition. However, also younger patients or parents can be overstrained with self-care demands. Recent research among the US population showed that poor health literacy is associated with more frequent healthcare utilization and expenditures, showing that poor health literacy also has impact on the healthcare system itself.

In this respect, adequate patient information is crucial. With every hospital visit - after hospitalisation or in the outpatient clinic - patients usually receive a referral letter which ideally describes the present symptoms or illness, the treatment carried out and steps the patient should take by herself/himself in the near or distant future. In reality these notes are often written in medical language that is difficult or impossible to understand for lays and usually contain information that is intended rather for communication between physicians or therapists. However, it is difficult to find a middle course that provides patients with adequate information while at the same time not losing informational content of immediate relevance for all professions involved in patient care.

Despite great efforts of all departments of the University Hospital Graz and all Styrian (KAGES) hospitals, adequate referral letters that also suffice the demands of stakeholders such as general practitioners, remains an issue needing further attention. Up to now, there has been no referral letter that provides both medical information for professionals as well as information that addresses the patient directly and is adapted to the respective medical knowledge.

Aim and Hypothesis The aim of this study is to develop and test an improved referral letter within the KAGES-wide project "Entlassungsdokumentation NEU"

ELIGIBILITY:
Inclusion Criteria:

* Patients of any department of the University Hospital Graz at the time of hospital discharge, or during waiting hours at the outpatient department (since those patients can be regarded as not critically ill and in a mental and physical state that will allow them to fill out a questionnaire).
* Physicians of any department of the University Hospital Graz and outside of the hospital, irrespective of their specialisation
* Nursing staff of any department of the University Hospital Graz and outside of the hospital, irrespective of the additional training
* Students of the Medical University of Graz, irrespective of the field of study

Exclusion Criteria:

* Patients who are critically ill and/or mentally or physically obviously not capable to partake in the survey
* Participants who are unwilling to partake, i.e. did not fill out the informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1000
Sampling Method: Non-Probability Sample
Enrollment: 982 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint of the study is the comprehension of medical content. | 1 day (single measurement by means of questionnaire)
  The comprehension of medical content is assessed with a questionnaire-based survey encompassing specific questions inquiring the understanding of medical information delivered in the referral letters. All questions are answered based on a Likert-scale. Improvement of comprehension will be measured via comparison of the results between the two groups.

SECONDARY OUTCOMES:
Subjective satisfaction with the referral letter | 1 day (single measurement by means of questionnaire)
  Subjective satisfaction is assessed with a questionnaire-based survey encompassing specific questions inquiring the understanding of medical information delivered in the referral letters. All questions are answered based on a Likert-scale. Improvement of comprehension will be measured via comparison of the results between the two groups.
Influence of demographic parameters on the understanding of medical content | 1 day (single measurement by means of questionnaire)
  The demographic parameters include age, gender, level of education and profession. The impact of demographic parameters will be measured by setting the survey results of both study groups into relation with age, gender, level of education or profession.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Smolle, Dr., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Schwarz CM, Hoffmann M, Smolle C, Borenich A, Furst S, Tuca AC, Holl AK, Gugatschka M, Grogger V, Kamolz LP, Sendlhofer G. Patient-centered discharge summaries to support safety and individual health literacy: a double-blind randomized controlled trial in Austria. BMC Health Serv Res. 2024 Jul 9;24(1):789. doi: 10.1186/s12913-024-11183-w. PMID 38982360